CLINICAL TRIAL: NCT03512145
Title: A Prospective Evaluation of the VIPUN Balloon Catheter 0.2: an Investigational Medical Device for the Monitoring of Gastric Motility in Adult Critically Ill Patients
Brief Title: Clinical Evaluation of the VIPUN Balloon Catheter 0.2 in Critically Ill Patients
Acronym: ANTERO-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Dr Jan Tack (Other)
Responsible Party: Sponsor-Investigator, Prof Dr Jan Tack, Member of staff hepato-gastroenterology, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S61147
Record Dates: First submitted 2018-03-30; First posted 2018-04-30 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Critical Illness; Intolerance; Nutritional; Delayed Gastric Emptying; Gastric Motor Dysfunction
MeSH Terms: conditions — Critical Illness; Gastroparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIPUN Balloon Catheter (Experimental): Recording of gastric motility with the investigational medical device. Gastric emptying rate of a liquid meal is assessed with the 13C-octanoate breath test.
  Interventions: Device: VIPUN Balloon Catheter

INTERVENTIONS:
Device: VIPUN Balloon Catheter — Gastric motility is recorded continuously with the VIPUN Balloon Catheter for 10 hours.

SUMMARY:
An open label, non-randomized, monocentric, interventional investigation in a cohort of adult critically ill patients

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Of adult age (18 years or older)
* ICU patients in which enteral nutrition is planned to be initiated and are expected to stay at least 1 day in ICU on enteral feeding.
* Patients should be mechanically ventilated or have an endotracheal tube or tracheostomy in place.

Exclusion Criteria:

* Contra-indication for (re-) placement of nasogastric feeding catheters.
* History of gastric or esophageal surgery
* Any gastrointestinal surgery or trauma that could significantly increase the risk related to the investigational medical device in the opinion of the investigator
* Fed by mouth or enterally prior to inclusion
* Patient is moribund
* Known pregnancy or breastfeeding women
* Receives gastroprokinetic medication (e.g., erythromycin, metoclopramide, domperidone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Gastric motility | 10 hours
  Assessed with the VIPUN Balloon Catheter
gastric emptying rate | 6 hours
  Assessed with 13C-octanoate breath test

SECONDARY OUTCOMES:
Success rate placement and removal balloon catheter | Day 0 until day 1 (<24 h)
  Success rate completing the procedures to place and remove the balloon catheter
Safety parameters potentially related to the use of the investigational medical device | Day 0 until day 30
  Incidence, frequency, severity, seriousness and relatedness of adverse events/effects are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No